CLINICAL TRIAL: NCT02648880
Title: The Effects of a Preoperative Exercise Intervention During Neoadjuvant Therapy in Patients With Pancreatic Cancer
Brief Title: Preoperative Exercise in Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-2266.cc
Record Dates: First submitted 2015-12-29; First posted 2016-01-07 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Cancer
Keywords: Exercise; Physical Activity
MeSH Terms: conditions — Pancreatic Neoplasms; Motor Activity | interventions — Resistance Training; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Group (Experimental): Participants will complete an exercise program in addition to standard care. Participants will start the exercise program within four weeks of their diagnosis and decision to undergo neoadjuvant treatment and continue until surgery. Participants will be encouraged to complete three sessions per week for at least eight weeks during neoadjuvant therapy. Exercise intensity, components, and time will be recorded for each exercise session. Participants will schedule their sessions with the exercise specialists administering the program, typically taking place between 8AM and 4PM, Monday through Friday.
  Interventions: Behavioral: Exercise program; Other: Standard Care
- Standard Care (Active Comparator): Participants in the Standard Care group will receive no exercise intervention, but will continue to receive standard follow-ups, treatments and services from their oncology team.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Exercise program — Individual exercise sessions in this program implement a "whole body" approach and consist of a 10-min cardiovascular warm-up and 50 minutes of cardiovascular endurance, resistance, and flexibility exercises. Target intensity of exercise will be based on the American College of Sports Medicine recommendations for cancer survivors. Prior to the start of exercise sessions, participants will be questioned on significant changes in symptoms or the presence of new symptoms (such as nausea or fever), which will used to modify the exercise session for that day to allow maximum symptom-limited participation.
  Arms: Exercise Group
Other: Standard Care — The services that participants receive as standard care include their medical care, symptom control, social worker support, and nutrition. These services are provided by their oncology team.

SUMMARY:
The purpose of this study is to investigate the effects of a preoperative exercise program in patients with pancreatic cancer preparing for surgery. Preoperative exercise programs have been shown to be effective in other cancer populations, but have not been investigated in patients with pancreatic cancer. The outcomes in this study will be changes in physical fitness, function, and postoperative outcomes. This investigation is a non-randomized control trial, with participants assigned to receive the preoperative exercise intervention in addition to standard care, or standard care alone if unable to commit to an exercise program for practical reasons. Possible mediators for the effects of exercise on postoperative outcomes will also be assessed, including psychological outcomes and markers of systemic inflammation. These measures will be assessed in all participants prior to program initiation, prior to surgery, and after surgery. Changes in these measures in response to exercise will be assessed, as well as the ability of the preoperative measures to predict postoperative outcomes.

DETAILED DESCRIPTION:
This study focuses on patients prescribed neoadjuvant (preoperative chemotherapy and radiation) prior to surgery for borderline resectable pancreatic adenocarcinoma. This allows for a known, preoperative window long enough to provide an effective exercise intervention. The exercise program will be administered for at least eight weeks, but has no cap on length, as neoadjuvent treatment periods can vary between participants and a cessation of the exercise program before the end of this period could result in an undesirable loss in physical fitness and function.

The study is a non-randomized, parallel group, intervention control trial, based on pilot studies in similar patient populations. All participants meeting the inclusion criteria and able to participate in the exercise program will be assigned to the exercise group. Participants meeting the inclusion criteria, but unable to commit to the exercise program for practical reasons (transportation, location, etc), will be assigned to the standard care group.

ELIGIBILITY:
Inclusion Criteria:

* Recent (< 4 week) first diagnosis of a borderline resectable pancreatic adenocarcinoma
* Prescription to receive neoadjuvant therapy and surgery,
* Age 21 to 80 years old,
* Physician clearance to participate in exercise program.

Exclusion Criteria:

* Any significant comorbid conditions that would interfere with or preclude participation in an exercise intervention, including orthopedic conditions such as advanced osteoarthritis, mobility-limiting amputations or chronic injuries, or mobility-limiting acute orthopedic injuries
* Advanced rheumatoid arthritis
* Widespread chronic pain conditions such as fibromyalgia
* Pulmonary conditions such as chronic obstructive pulmonary disease, emphysema, interstitial lung disease, use of supplementary oxygen
* Known cardiovascular disease or new cardiac event in last 6 months
* Diabetes
* Pregnancy
* Second cancer diagnosis at the time of enrollment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Jankowski, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Health and Wellness Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
This is a small, non-FDA Regulated pilot study of an exercise intervention.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Group
Started | 3 (Recruitment was significantly limited, only 3 participants were eligible, all enrolled. All three were assigned to the exercise arm, per protocol. No participants were recruited into the control arm and it was eliminated.)
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exercise Group
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in 400-meter Walk Time
Description: Assessment of physical fitness and function. Participants are timed while walking 400 meters at a fast, but safe, pace.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Population: One participant did not receive surgery and was excluded from the postoperative timepoint.
Measure: Mean (Full Range); unit: s
Arm/Group | Exercise Group
Number analyzed (Participants) | 3
s
  Baseline | 212.7 [211 to 214]
  Pre-operative | 194.3 [188 to 205]
  Postoperative: number analyzed (Participants) | 2
  Postoperative | 204 [195 to 213]

2. Secondary Outcome: Change in Body Composition
Description: Assessment of physical fitness. Dual-energy x-ray absorptiometry (DXA) will assess lean muscle mass and body fat.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

3. Secondary Outcome: Change in Gait Speed
Description: Participant gait speed will be determined on a 10 meter course for both fast and self-selected paces.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

4. Secondary Outcome: Change in Timed Up and Go
Description: Participants are timed as they rise from a chair, walk 3 meters, turn around, and return to the chair and sit.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

5. Secondary Outcome: Change in Stair Climb Test
Description: Participants are timed as they ascend and descend one flight of stairs.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

6. Secondary Outcome: Change in Single Limb Stance
Description: Participants are timed on how long they can balance on one leg.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

7. Secondary Outcome: Change in 30 Second Sit-to-Stand
Description: The number of times a participant can rise from a chair in 30 seconds is counted.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

8. Secondary Outcome: Change in Grip Strength
Description: The maximum force the participant can produce separately with both hands, assessed by grip dynamometry, is measured.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

9. Secondary Outcome: Change in Average Daily Step Count
Description: The average step count for a minimum of 3 days over a 7 day period will be assessed with accelerometry.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

10. Secondary Outcome: Change in Wellness
Description: The Colorado Comprehensive Wellness Assessment, a survey, will be administered to assess eight domains of wellness.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

11. Secondary Outcome: Change in Health-related Quality of Life
Description: The Functional Assessment of Cancer Therapy - General Form (FACT-G), a survey, will be administered.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

12. Secondary Outcome: Change in Perceived Fatigue
Description: Perceived fatigue will be assessed by the Revised Piper Fatigue Scale, a survey.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

13. Secondary Outcome: Change in Anxiety
Description: Changes in state and trait anxiety will be assessed with the Spielberger State-Trait Anxiety Index.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

14. Secondary Outcome: Change in Perceived Stress
Description: Changes in perceived stress will be assessed with the Perceived Stress Scale.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

15. Secondary Outcome: Resting Heart Rate Variability
Description: Heart rate variability will be assessed from electrocardiography (ECG) obtained during a 5 min rest period.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

16. Secondary Outcome: Heart Rate Variability Response to Physiologic Challenge
Description: Heart rate variability will be assessed from electrocardiography (ECG) obtained during a 5 min rest period, and changes in response to a physiologic challenge (orthostatic stress: chair rise).
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

17. Secondary Outcome: Heart Rate Variability Response to Mental Stressor
Description: Heart rate variability will be assessed from electrocardiography (ECG) obtained during a 5 min rest period, and changes in response to a mental challenge (Stroop Task).
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

18. Secondary Outcome: Heart Rate Variability Response to a Cancer-specific Mental Stressor
Description: Heart rate variability will be assessed from electrocardiography (ECG) obtained during a 5 min rest period, and changes in response to a cancer-specific mental challenge (Cancer-Specific Stroop Task).
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

19. Secondary Outcome: Change in C-reactive Protein
Description: Serum C-reactive protein will be assessed from blood draws.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

20. Secondary Outcome: Change in Interleukin-6
Description: Serum interleukin-6 will be assessed from blood draws.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

21. Secondary Outcome: Change in Soluble Tumor-necrosis Factor Receptor 1
Description: Soluble tumor-necrosis factor receptor 1 will be assessed from blood draws.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

22. Secondary Outcome: Change in Interleukin-10
Description: Serum interleukin-10 will be assessed from blood draws.
Time Frame: Baseline, Pre-operative (within the 2 weeks prior to surgery), 6 weeks postoperative
Reporting Status: Not Posted

23. Secondary Outcome: Determination of Hospital Length of Stay
Description: At 30 days after discharge from the hospital, a medical record review will be conducted to determine the number of days participants were in the hospital after surgery.
Time Frame: 30 days after hospital discharge
Reporting Status: Not Posted

24. Secondary Outcome: Determination of Hospital Readmission
Description: At 30 days after discharge from the hospital, a medical record review will be conducted to determine whether participants were readmitted to the hospital for an unplanned surgical complication in the 30 days following hospital discharge.
Time Frame: 30 days after hospital discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 6 months. From baseline assessment through 6 weeks after surgery.
Arm/Group | Exercise Group
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02648880/Prot_SAP_ICF_000.pdf